CLINICAL TRIAL: NCT01841541
Title: Triage Plus for TB: Improving Community-Based Provision for TB in Africa. The Impact of Involving Informal Health Providers for Tuberculosis Control in Sudan
Brief Title: The Impact of Involving Informal Health Providers for Tuberculosis Control in Sudan
Acronym: Triage-Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: The Epidemiological Laboratory (EpiLab), Khartoum-Sudan. (Unknown); The Norwegian Heart and Lung Patients Association (LHL) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11.03RS
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Informal providers; Informal carers; Barriers to health system
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ombda Locality: informal providers (Experimental): Ombda locality is located in Western Khartoum and populated with population size of 988,163.
  Intervention: 380 unpaid Informal providers trained to recognise TB symptoms and to refer presumptive TB cases to formal health care facilities within the area.
  Interventions: Behavioral: Referral of presumptive of TB cases by informal providers
- Jabal Awlia Locality (No Intervention): The control arm: A locality in south eastern site of Khartoum state populated with 942,429. No intervention took place

INTERVENTIONS:
Behavioral: Referral of presumptive of TB cases by informal providers — Training of informal providers to effectively refer TB suspects in the community to the primary health care system
  Arms: Ombda Locality: informal providers

SUMMARY:
Training and engaging of unpaid informal providers (such as tea-sellers, women's groups, youth clubs, small traders and religious groups) from poorer localities in TB disease recognition, referral and community awareness raising will increase the access of TB patients to formal health facilities and decrease their delay in initiating TB treatment.

DETAILED DESCRIPTION:
Barriers to accessing health services faced by poor and vulnerable populations are numerous in developing countries. These include; geography, income poverty, lack of trust in the quality of public health services, and lack of empowerment of women and adolescent girls (as patients and carers) to mobilize adequate and timely resources to access these services.

The project aims to test if TB case detection can be increased by engaging informal health care providers in active case finding. In one urban district of Khartoum, these providers will be trained to work as first point of entry to the health system using a comprehensive package that includes disease recognition, health communication, and patient referral. In a comparator urban district of Khartoum, no attempts will be made to engage informal providers.

By comparing data of TB patients and Lab registers between the intervention and comparator districts in Khartoum, this project aims to test if, and to what extent, these expected effects can be realized.

Overall this is a trial of a health policy so individual patients will not be recruited or randomized to one intervention or the other. Rather the policy is being applied in one district while the other district is being used as a comparator.

ELIGIBILITY:
Inclusion Criteria:

* Access point for health seeking by the poor and vulnerable
* Active and well known in community
* Intervention activities can be confined to intervention area
* Based in community/locality
* Longevity; long standing
* Present in control and intervention areas
* Able and willing to complete the training to be Triage-Plus providers (ie giving formal consent)

Exclusion Criteria:

* Formal health providers, e.g. clinics, labs, hospitals (MOH, NGO or private)
* Internationally funded organizations, e.g. international NGOs
* Civil servants e.g. teachers

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Total number of TB patients registered and start receiving treatment in formal health care facilities | 12 months
  This will be measured by comparing Data from routine patients registered in formal TB management units in the intervention arm and compare it with the same routine data from the control arm. similar data for the previous year will undergo the same comparison as time control for both arms

CONTACTS AND LOCATIONS:
Overall Officials: S. Bertel ("Bertie") Squire, MB BChir, MD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- The Epidemiological Laboratory (EpiLab), Khartoum, Khartoum State, Sudan